CLINICAL TRIAL: NCT02087111
Title: Telaprevir in Patients With Genotype 3 HCV: Pilot Clinical Study to Evaluate Efficacy and Predictability of Therapy in Patients Who Have Failed to Respond to Pegylated Interferon and Ribavirin
Brief Title: Telaprevir in Genotype 3 HCV
Acronym: TIG3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Barts & The London NHS Trust (Other); St George's Healthcare NHS Trust (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9132; 2013-003729-27 (EudraCT Number); 13/LO/1473 (Other: Health Research Authority)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: Telaprevir; Genotype 3 HCV
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): All patients who are fulfil the entry criteria are treated for 24 weeks with 40 Kd Pegylated interferon alfa 2a, Ribavirin and 12 weeks with telaprevir.
  Interventions: Drug: Telaprevir; Drug: 40 Kd Pegylated interferon alfa 2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — 375 mg film coated tablets
  Other Names: INCIVO
Drug: 40 Kd Pegylated interferon alfa 2a — 180 µg in pre-filled syringe for sub-cutaneous injection
  Other Names: Pegasys
Drug: Ribavirin — 200 mg tablets
  Other Names: Copegus

SUMMARY:
Patients with genotype 3 hepatitis C who have advanced liver disease (cirrhosis) have a very high chance of developing fatal complications of their disease unless they receive effective treatment. Unfortunately the best drugs that are currently available to treat genotype 3 hepatitis C (pegylated interferon and ribavirin) only work in about 50% of patients with advanced liver disease and therefore a large number of patients who have failed treatment are waiting for new, better drugs. Currently there are no treatments available for these patients. Telaprevir is a new drug that is licensed to treat genotype 1 hepatitis C and which works very well in these patients. In patients with genotype 3 hepatitis C small scale trials and laboratory studies show that some patients do respond quite well and others respond a little bit when given telaprevir. In patients who have exhausted all other treatment options the investigators speculate that telaprevir treatment may help some patients by clearing their infection. The purpose of this study is to see if telaprevir can help these patients and to determine if the investigators can predict in advance which people can be helped.

DETAILED DESCRIPTION:
This is an open label, 'proof of concept' study to examine the hypothesis that telaprevir is effective in patients with genotype 3 HCV and cirrhosis who have failed to respond to pegylated interferon and ribavirin. The study will examine the hypothesis that pretreatment viral testing will identify patients who will respond to antiviral therapy with telaprevir.

Patients who are eligible for the study will be asked if they are willing to participate and if they wish to join the study they will be asked to sign the informed consent form. After signing the consent form patients will attend the hospital and be screened for the trial. This will involve a physical examination and blood samples will be taken. Patients will be provided with an injection of pegylated interferon to be self administered every week along with ribavirin tablets (4 tablets a day) and telaprevir tablets (6 tablets a day). Patients will be taught how to self administer the pegylated interferon medication. Patients will reattend every week for the next 4 weeks. At each visit they will be asked questions about the medication that they are taking, questions about how they are feeling and any side effects and 30 mls of blood will be taken.

At the fourth visit (week 4) the amount of circulating HCV will be assessed using a standard laboratory assay and patients will be telephoned within 1 week of the visit. If the viral load is more than 1000 IU/ml therapy will be stopped as the chance of the patient responding to therapy is very low (in the clinical studies with genotype 1 HCV no patients responded who had a viral load of >1000 IU/ml at week 4). If patients are responding to therapy they will be asked to continue with medication and seen again 4 weeks later (8 weeks after initiating therapy).

At week 8 of therapy patients will be asked questions about the medication that they are taking, questions about how they are feeling and any side effects and blood will be taken. Again the viral load will be tested and if the viral load is more than 1000 IU/ml therapy or the viral load has not decreased by 3 logs from baseline therapy will be stopped as the chance of the patient responding to therapy is very low. If patients are responding to therapy they will be asked to continue with medication and seen again 4 weeks later (12 weeks after initiating therapy).

At week 12 of therapy patients will be asked questions about the medication that they are taking, questions about how they are feeling and any side effects and blood will be taken. At this visit they will be told to stop taking the telaprevir tablets as the recommended duration of telaprevir therapy is 12 weeks. Patients will continue to take pegylated interferon and ribavirin.

Patients will be seen again every 4 weeks for another 8 weeks and they will continue to take pegylated interferon injections every week and 4 ribavirin tablets every day. At each clinic visit they will be asked questions about the medication that they are taking, questions about how they are feeling and any side effects and blood will be taken.

After 24 weeks of therapy (i.e. 4 weeks after the last visit) patients will be seen again and asked questions about the medication that they are taking, questions about how they are feeling and any side effects and blood will be taken. At this visit they will be told to stop taking all medication. They will be asked to return in 12 weeks.

12 weeks after stopping therapy patients will return to the clinic and asked questions about how they are feeling and any side effects and blood will be taken. They will be asked to return in 12 weeks.

24 weeks after stopping therapy patients will return to the clinic and asked questions about how they are feeling and any side effects and blood will be taken. The study will then end and they will return to routine clinical follow up where they will be seen by their clinical team.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years of age and ≤ 70 years old
* Advanced fibrosis - defined as a liver biopsy within 2 years showing an Ishak fibrosis score of >4 OR radiological evidence of cirrhosis (ultrasound scan or fibroscan reading >10.6)
* Previous therapy with pegylated interferon and ribavirin for at least 24 weeks with undetectable HCV RNA at the end of therapy and detectable HCV RNA six months after treatment cessation
* Chronic genotype 3 HCV infection, RNA positivity with genotype 3 infection confirmed at a local laboratory.
* HBsAg negative and no clinical evidence of co-infection with HIV
* Platelet count >50,000 cells/mm3 (support with eltrombopag is permitted) Neutrophil count > 600 cells/mm3
* All female patients of childbearing potential and all males with female partners of childbearing potential must be prepared to use two forms of effective contraception* (combined) during treatment and 6 months after treatment end
* Able and willing to give informed consent and able to comply with study requirements

Exclusion Criteria:

* Evidence of other cause of significant liver disease - serum ferritin > 1000, biochemical evidence of Wilson's disease, autoantibody titres in excess of 1:160
* Poorly controlled diabetes that, in the investigators opinion, precludes therapy
* Severe retinopathy that, in the opinion of the investigator, precludes therapy
* Evidence of ascites seen on previous liver ultrasound
* Haemoglobin concentration <11 g/dL in females or <12 g/dL in males or any patient with an increased risk for anaemia (e.g., thalassemia, sickle cell anaemia, spherocytosis, history of gastrointestinal bleeding) or for whom anaemia would be medically problematic
* Albumin levels <35 G/L
* Females who are pregnant or breast-feeding
* History of severe psychiatric disease, including psychosis and/or depression, characterized by a suicide attempt, hospitalization for psychiatric disease, or a period of disability as a result of psychiatric disease within the last 2 years
* History of immunologically mediated disease (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune haemolytic anaemia, scleroderma, severe psoriasis (defined as affecting >10% of the body, where the palm of one hand equals 1%, or if the hands and feet are affected), rheumatoid arthritis requiring more than intermittent nonsteroidal anti-inflammatory medications for management
* Other on-going serious medical condition in the opinion of the investigator that would prohibit treatment
* Poorly controlled thyroid dysfunction that, in the investigators opinion, precludes therapy
* History of major organ transplantation with an existing functional graft
* History of severe pre-existing cardiac disease, including unstable or uncontrolled cardiac disease in the previous 6 months
* History or laboratory testing showing evidence of a haemoglobinopathy
* Concomitant administration with active substances that are highly dependent on CYP3A for clearance and for which elevated plasma concentrations are associated with serious and/or life-threatening events. These active substances include alfuzosin, amiodarone, bepridil, quinidine, astemizole, terfenadine, cisapride, pimozide, ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine), lovastatin, simvastatin, atorvastatin, sildenafil or tadalafil (only when used for treatment of pulmonary arterial hypertension) and orally administered midazolam or triazolam.
* Concomitant administration with Class Ia or III antiarrhythmics, except for intravenous lidocaine (see section 4.5).
* Concomitant administration of INCIVO with active substances that strongly induce CYP3A e.g. rifampicin, St John's wort (Hypericum perforatum), carbamazepine, phenytoin and phenobarbital and thus may lead to lower exposure and loss of efficacy of INCIVO.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) 12 weeks after end of treatment (SVR12) | Week 36
  To determine whether patients with genotype 3 HCV and cirrhosis who have relapsed following therapy with PegIFN and RBV will achieve a sustained virological response (SVR) if treated with telaprevir, PegIFN and RBV

SECONDARY OUTCOMES:
Response rate prediction | By week 12
  The proportion of patients who are phenotypically poorly responsive to telaprevir (defined as virus with a poor response to telaprevir in vitro i.e. an IC50 of <0.1microMol in an in vitro assay) who achieve early and late virological clearance.
Sustained virological response 24 weeks after end of treatment. | week 48
  The proportion of patients with a sustained virological response 24 weeks after the last dose of PegIFN and RBV (SVR24). SVR 24 is defined as undetectable HCV RNA on a blood sample taken between 24 and 30 weeks after the final dose of PegIFN and ribavirin measured using a sensitive, validated polymerase chain reaction (PCR) assay with a lower limit of quantification of at least 30IU/ml.
Treatment Success | After week 48
  The proportion of patients who have undetectable HCV RNA (measured using a sensitive, validated polymerase chain reaction (PCR) assay with a lower limit of quantification of at least 30IU/ml) after 1,2,3 and 4 weeks of therapy with PegIFN, RBV and telaprevir.

CONTACTS AND LOCATIONS:
Overall Officials: Graham R Foster, Principal Investigator — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Barts Health NHS Trust, London
  - Ste Georges Healthcare NHS Trust, London
  - Nottingham University Hospitals Trust, Nottingham

REFERENCES:
- [Background] Shoeb D, Rowe IA, Freshwater D, Mutimer D, Brown A, Moreea S, Sood R, Marley R, Sabin CA, Foster GR. Response to antiviral therapy in patients with genotype 3 chronic hepatitis C: fibrosis but not race encourages relapse. Eur J Gastroenterol Hepatol. 2011 Sep;23(9):747-53. doi: 10.1097/MEG.0b013e3283488aba. PMID 21691208
- [Background] Alazawi W, Cunningham M, Dearden J, Foster GR. Systematic review: outcome of compensated cirrhosis due to chronic hepatitis C infection. Aliment Pharmacol Ther. 2010 Aug;32(3):344-55. doi: 10.1111/j.1365-2036.2010.04370.x. Epub 2010 May 22. PMID 20497143
- [Background] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307
- [Background] Zeuzem S, Andreone P, Pol S, Lawitz E, Diago M, Roberts S, Focaccia R, Younossi Z, Foster GR, Horban A, Ferenci P, Nevens F, Mullhaupt B, Pockros P, Terg R, Shouval D, van Hoek B, Weiland O, Van Heeswijk R, De Meyer S, Luo D, Boogaerts G, Polo R, Picchio G, Beumont M; REALIZE Study Team. Telaprevir for retreatment of HCV infection. N Engl J Med. 2011 Jun 23;364(25):2417-28. doi: 10.1056/NEJMoa1013086. PMID 21696308
- [Background] Foster GR, Hezode C, Bronowicki JP, Carosi G, Weiland O, Verlinden L, van Heeswijk R, van Baelen B, Picchio G, Beumont M. Telaprevir alone or with peginterferon and ribavirin reduces HCV RNA in patients with chronic genotype 2 but not genotype 3 infections. Gastroenterology. 2011 Sep;141(3):881-889.e1. doi: 10.1053/j.gastro.2011.05.046. Epub 2011 May 31. PMID 21699786